CLINICAL TRIAL: NCT04269915
Title: Establishing a Female-only Controlled Human Schistosoma Mansoni Infection Model: a Safety and Dose Finding Study (CoHSI2)
Brief Title: Single-sex Female Controlled Human Schistosomiasis Mansoni Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CoHSI2
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Schistosomiasis; Schistosomiasis Mansoni
MeSH Terms: conditions — Schistosomiasis; Schistosomiasis mansoni

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Volunteers will be exposed to escalating doses of female Schistosoma mansoni cercariae
  Interventions: Biological: female Schistosoma mansoni cercariae

INTERVENTIONS:
Biological: female Schistosoma mansoni cercariae — Viable female Schistosoma mansoni cercariae of the Puerto Rican strain

SUMMARY:
Groups of 3 or 7 volunteers will be exposed to a predetermined number of female Schistosoma mansoni cercariae until 10 volunteers are found infected.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 18 and ≤ 45 years and in good health.
* Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
* Subject is able to communicate well with the investigator, is available to attend all study visits.
* Subject will remain within Europe (excluding Corsica) during the study period and is reachable by mobile telephone from week 3 to week 8 of the study period.
* Subject agrees to refrain from blood donation to "Sanquin" (blood bank) or for other purposes throughout the study period.
* For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
* Subject has signed informed consent.

Exclusion Criteria:

* Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

  * body weight <50 kg or Body Mass Index (BMI) <18.0 or >30.0 kg/m2 at screening;
  * positive human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) screening tests;
  * the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period;
  * history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years;
  * any history of treatment for severe psychiatric disease by a psychiatrist in the past year;
  * history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
  * The chronic use of any drug known to interact with praziquantel, artesunate or lumefantrine metabolism (e.g. phenytoin, carbamazepine, phenobarbital, primidon, dexamethasone, rifampicin, cimetidine, flecainide, metoprolol, imipramine, amitriptyline, clomipramine, class I-A and III anti-arrythmics, antipsychotics, antidepressants, macrolides, fluoroquinolones, imidazole- and triazole antimycotics, antihistamines) Because lumefantrine may cause extension of QT-time, chronic use of drugs with effect on QT interval are excluded from the study.
* For female subjects: positive urine pregnancy test at screening.
* Any history of schistosomiasis or treatment for schistosomiasis.
* Positive serology for schistosomiasis or elevated serum CAA at screening.
* Known hypersensitivity to or contra-indications (including co-medication) for use of praziquantel, artesunate or lumefantrine.
* Being an employee or student of the department of parasitology or infectious diseases of the Leiden University Medical Center.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events, possibly, probably or definitely related to controlled human Schistosoma mansoni infection with female cercariae. | 20 weeks
Number of female cercariae at which 100% volunteers show detectable Schistosoma mansoni circulating anodic antigen. | 8 weeks

SECONDARY OUTCOMES:
Average number of weeks until positive serum circulating anodic antigen (CAA) test | 8 weeks
Comparison of peak serum circulating anodic antigen (CAA) concentration in different dose groups | 8 weeks
Humoral (antibody) response profile by protein and glycan array between infected and uninfected individuals | 1 year
Ex vivo lymphocyte profiles using flow cytometry between infected and uninfected individuals | 1 year
Changes over time in commensal gut bacteria by looking at the relative abundance of microbiota using 16S rRNA gene amplicon sequencing after controlled human Schistosoma mansoni infection with female cercariae | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koopman JPR, Houlder EL, Janse JJ, Casacuberta-Partal M, Lamers OAC, Sijtsma JC, de Dood C, Hilt ST, Ozir-Fazalalikhan A, Kuiper VP, Roozen GVT, de Bes-Roeleveld LM, Kruize YCM, Wammes LJ, Smits HH, van Lieshout L, van Dam GJ, van Amerongen-Westra IM, Meij P, Corstjens PLAM, Jochems SP, van Diepen A, Yazdanbakhsh M, Hokke CH, Roestenberg M. Safety and infectivity of female cercariae in Schistosoma-naive, healthy participants: a controlled human Schistosoma mansoni infection study. EBioMedicine. 2023 Nov;97:104832. doi: 10.1016/j.ebiom.2023.104832. Epub 2023 Oct 12. PMID 37837930